CLINICAL TRIAL: NCT01181882
Title: The Effects of Fish Oil and Aspirin on Cardiovascular Risk in Type 2 Diabetes
Brief Title: Fish Oil and Aspirin With Type 2 Diabetes
Acronym: R-21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Cornell University (Other); Albany College of Pharmacy and Health Sciences (Other)
Responsible Party: Principal Investigator, Robert Block, Assistant Professor, University of Rochester
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: RSRB00030668
Record Dates: First submitted 2010-08-03; First posted 2010-08-13 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease; Aspirin Resistance; Diabetes Mellitus, Type 2; Platelet Function; Omega-3 Fatty Acids; Aspirin; Lysophospholipids; Lysophosphatidic Acid; Lysophosphatidylcholine
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — Fish Oils; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fish Oil and Aspirin (Experimental)
  Interventions: Dietary Supplement: Fish Oil and Aspirin

INTERVENTIONS:
Dietary Supplement: Fish Oil and Aspirin — 4 grams of fish oil each day for 28 days and 81 mg aspirin
  Other Names: Omega-3 EPA/DHA Concentrate; Aspirin

SUMMARY:
The purpose of this study is to understand if omega-3 fatty acids in fish oil enhance the ability of aspirin to reduce the risk of cardiovascular diseases such as heart attack and stroke in those who have diabetes mellitus.

DETAILED DESCRIPTION:
A recent increase in the incidence and prevalence of obesity-related diabetes mellitus and the metabolic syndrome as a result of insulin resistance threatens to reverse the health gains achieved in the US during the last half of the 20th century. Novel inexpensive and safe pharmacologic approaches are required to prevent a variety of resulting cardiovascular disease sequelae. Aspirin is a proven agent in the treatment and prevention of cardiovascular disease but is greatly underused. Even when it is used, aspirin is ineffective in a large proportion of the population: a problem termed "aspirin resistance." Approximately thirty percent of the adult US population is aspirin resistant and this proportion is higher in those with diabetes and the metabolic events and affected patients do not benefit from other antiplatelet drugs. The omega-3 fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are naturally occurring and can be safely used at low cost in individuals who are in high and lower cardiovascular risk groups. Supplementation with EPA and and DHA (EPA + DHA) modifies the fatty acid balance which is distributed in patients with insulin resistance and atherosclerosis, thereby potentially improving endothelial function, lowering blood pressure, and reducing the risk of fatal and non-fatal acute coronary syndromes. Emerging evidence indicates that the combination of aspirin together with EPA+DHA supplementation beneficially regulates fatty acid metabolism and attenuates atherosclerosis. However, the effects of aspirin together with EPA + DHA on aspirin resistance or in subjects with diabetes mellitus and insulin resistance are unknown. Circulating EPA and DHA are contained largely in lysophospholipids, which contain a three carbon backbone and variable fatty acyl side chains. In preliminary data, we show that both aspirin ingestion and EPA+DHA supplementation after lysophospholipids including lysophosphatidylcholine (LPC) and lysophosphatidic acid (LPA) are now known to bind specific G-protein coupled receptors, which are being explored as novel therapeutic targets in cardiovascular and other diseases. Relationships between LPC and LPA metabolism, aspirin ingestion, and human atherosclerosis have not been investigated (to our knowledge). In the proposed study, we will investigate the effects of combining aspirin with EPA+DHA supplementation on platelet function and lysophospholipid metabolism in a clinical trial of individuals with type 2 diabetes mellitus. This trial will build on existing infrastructure in clinical and translational research, as well as our preliminary data using novel in-house assays.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40-80
* No significant abnormality noted from the CBC, CMP, TSH
* Have diabetes mellitus based on the criteria from the Report of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. (57) These data will be collected from medical records in conjunction with the Greater Rochester Practice-Based Research Network (see recruitment plan below)

  1. Symptoms of diabetes plus casual plasma glucose concentration greater than or equal to 200 mg/dl (11.1 mmol/l). Casual is defined as any time of day without regard to last time since last meal. The classic symptoms of diabetes include polyuria, polydipsia, and unexplained weight loss, or;
  2. Fasting plasma glucose greater than or equal to 126 mg/dl (11.1 mmol/l). Fasting is defined as no caloric intake for at least 8 h, or;
  3. 2-hour plasma glucose greater than or equal to 200 mg/dl (11.1 mmol/l) during an oral glucose tolerance test. The test should be performed as described by the World Health organization, using a glucose load containing the equivalent of 75 g anhydrous glucose dissolved in water. This is the protocol within the University of Rochester Clinical Labs.

(In the absence of unequivocal hyperglycemia with acute metabolic decompensation, these criteria should have been confirmed by repeat testing on a different day)

* Available for two morning visits (5 hours at bedrest) approximately 28 days apart and 2 short visits for blood draws
* No fish oil, flax seed oil, vitamins, nutri. supplements or herbal preps. during study
* Able to commit to no aspirin, NSAIDS for 10 days prior to each 5-hour study visit
* Able to commit to no more then 2 meals of fish 7 days prior to each visit
* Non-smoker
* Not currently pregnant, and will not become pregnant during study

Exclusion Criteria:

* History of drug or alcohol abuse, or current weekly alcohol consumption >14 units/week (1 unit=1 beer, 1 glass of wine, 1 mixed cocktail containing 1 ounce of alcohol)
* Diagnosis of cardiovascular disease including coronary heart disease, congestive heart failure, peripheral vascular disease, stroke, atrial fibrillation, and gastric bypass surgery or malabsorption syndrome.
* History of malignancy (unless disease free for >10 years, or non-melanoma skin carcinoma)
* History of peptic ulcer or gastrointestinal bleeding in past 5 years
* Diagnosed bleeding disorder
* Use of antiplatelet or antithrombotic therapy, defined as clopidogrel, ticlopidine, cilostazol, dipyridamol, trapidil, warfarin, and argatroban

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Platelet function | 4 hours
  Platelet function effect will be measured with aspirin alone and 4 hours later, after fish oil ingestion.

SECONDARY OUTCOMES:
Lysophospholipids | 4 hours
  Plasma measurement of lysophospholipids will be measured with aspirin alone and 4 hours later, after fish oil ingestion. These analyses will be considered exploratory due to the fact that no previous data exist regarding the relationships investigated and multiple testing is inherent to these analyses as 11 species of each LPA and LPC will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Block, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- Clinical Research Center of the University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Derived] Block RC, Abdolahi A, Tu X, Georas SN, Brenna JT, Phipps RP, Lawrence P, Mousa SA. The effects of aspirin on platelet function and lysophosphatidic acids depend on plasma concentrations of EPA and DHA. Prostaglandins Leukot Essent Fatty Acids. 2015 May;96:17-24. doi: 10.1016/j.plefa.2014.12.005. Epub 2014 Dec 22. PMID 25555354
- [Derived] Abdolahi A, Georas SN, Brenna JT, Cai X, Thevenet-Morrison K, Phipps RP, Lawrence P, Mousa SA, Block RC. The effects of aspirin and fish oil consumption on lysophosphatidylcholines and lysophosphatidic acids and their correlates with platelet aggregation in adults with diabetes mellitus. Prostaglandins Leukot Essent Fatty Acids. 2014 Feb-Mar;90(2-3):61-8. doi: 10.1016/j.plefa.2013.12.004. Epub 2013 Dec 18. PMID 24373610
- [Derived] Block RC, Abdolahi A, Smith B, Meednu N, Thevenet-Morrison K, Cai X, Cui H, Mousa S, Brenna JT, Georas S. Effects of low-dose aspirin and fish oil on platelet function and NF-kappaB in adults with diabetes mellitus. Prostaglandins Leukot Essent Fatty Acids. 2013 Jul;89(1):9-18. doi: 10.1016/j.plefa.2013.03.005. Epub 2013 May 7. PMID 23664596